CLINICAL TRIAL: NCT00945451
Title: Study of Doses Escalation on Efficacy on Cyberknife After Docetaxel-Cisplatin Concomitant Radiotherapy for Non Small Cells Lung Cancer Stage III
Brief Title: Stereotactic Radiosurgery in Treating Patients Undergoing Chemotherapy and Radiation Therapy For Stage III Non-Small Cell Lung Cancer
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Antoine Lacassagne (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CDR0000639362; CALACASS-CYBERTAXCIS; INCA-RECF0941; 2008-A01104-51
Record Dates: First submitted 2009-07-23; First posted 2009-07-24 (Estimated); Last update posted 2019-09-16 (Actual); Status verified 2018-02

CONDITIONS: Lung Cancer
Keywords: stage IIIA non-small cell lung cancer; stage IIIB non-small cell lung cancer; stage II non-small cell lung cancer
MeSH Terms: conditions — Lung Neoplasms; Carcinoma, Non-Small-Cell Lung

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- CyberKnife irradiation (Experimental)
  Interventions: Device: CK

INTERVENTIONS:
Device: CK — Cyberknife Irradiation

SUMMARY:
RATIONALE: Drugs used in chemotherapy, such as docetaxel and cisplatin, work in different ways to stop the growth of tumor cells, either by killing the cells or by stopping them from dividing. Stereotactic radiosurgery can send x-rays directly to the tumor and cause less damage to normal tissue. Giving stereotactic radiosurgery after docetaxel and cisplatin may kill more tumor cells.

PURPOSE: This phase I/II trial is studying the side effects and the best dose of stereotactic radiosurgery when given after docetaxel, cisplatin, and radiation therapy and to see how well it works in treating patients with stage III non-small cell lung cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* Evaluate the maximum tolerated dose of stereotactic radiosurgery in patients with locally advanced non-small cell lung cancer undergoing concurrent chemoradiotherapy. (Phase I)
* Assess the response rate (complete and partial response) in these patients by RECIST criteria. (Phase II)

Secondary

* Determine the tolerability. (Phase I)
* Assess the quality of life of these patients by QLQ-C30 v3. (Phase I)
* Assess the overall and disease-free survival of these patients. (Phase II)
* Assess progression-free survival of these patients. (Phase II)

OUTLINE: This is a multicenter, phase I dose escalation study of stereotactic radiosurgery followed by a phase II study.

Patients receive docetaxel IV and cisplatin IV on days 1, 22, 43, 50, 57, and 64 in the absence of disease progression or unacceptable toxicity. Beginning on day 43, patients undergo concurrent radiotherapy to the mediastinum 5 days a week. Beginning 2-3 weeks after chemoradiotherapy, patients undergo stereotactic radiosurgery on days 1, 3, and 5.

Quality of life is assessed by the QLQ-C30 v3 questionnaire at baseline, after radiosurgery, and at 6 and 12 months after completion of study treatment.

After completion of study treatment, patients are followed up monthly for 6 months, every 3 months for 1 year, and then every 6 months for 3 years.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed non-small cell lung cancer

  * Locally advanced disease
* No metastatic disease
* Unable to undergo surgery after concurrent chemoradiotherapy
* Must have 1-3 tumor target masses < 5 cm in greatest diameter and separated by ≥ 2 cm after concurrent chemoradiotherapy

PATIENT CHARACTERISTICS:

* WHO performance status 0-2
* Platelet count > 100,000/mm³
* Hemoglobin > 9 g/dL
* Neutrophil > 1.0 x 10^9/L
* FEV_1 > 30% of vital capacity
* Vital capacity > 25% of predicted value
* DLCO > 25% of predicted value
* LVEF ≥ 35%
* PT > 80
* aPTT > 35 sec
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception during and for 6 months after completion of study treatment
* Not under guardianship
* No dyspnea related to NYHA class III-IV heart failure
* No indirect signs of pulmonary arterial hypertension (pulmonary arterial systolic BP > 45 mm Hg)
* No pulmonary acceleration time < 100 ms
* No contraindication to fiducial insertion
* No geographical, social, or psychological conditions that would interfere with medical follow-up

PRIOR CONCURRENT THERAPY:

* Docetaxel and platinum-based drugs with concurrent irradiation allowed
* No prior surgery or surgery after the first phase of treatment with concurrent chemoradiotherapy
* No prior irradiation to lung
* No concurrent participation in another study trial

Ages: 18 Years to 120 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 35 (Actual)
Dates: Start 2009-04-24 (Actual); Primary Completion 2016-11-17 (Actual); Study Completion 2016-11-17 (Actual)

PRIMARY OUTCOMES:
Maximum tolerated dose (phase I) | 5 years
Overall response rate by RECIST (phase II) | 5 years

CONTACTS AND LOCATIONS:
Overall Officials: Pierre-Yves Bondiau, MD, PhD, Principal Investigator — Centre Antoine Lacassagne
Locations (1):
- Centre Antoine Lacassagne, Nice, France